CLINICAL TRIAL: NCT00006351
Title: Phase II Study on SCH 66336 (Farnesyl Protein Transferase Inhibitor) and Gemcitabine as Second Line Treatment in Advanced Metastatic Urothelial Cancer - EORTC Study 16997
Brief Title: SCH 66336 Plus Gemcitabine in Treating Patients With Advanced Cancer of the Urinary Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16997; EORTC-16997; EORTC-GU-16997; EORTC-PAMM-16997
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; recurrent urethral cancer; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Gemcitabine; lonafarnib

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: lonafarnib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining SCH 66336 and gemcitabine may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of SCH 66336 plus gemcitabine in treating patients who have advanced cancer of the urinary tract.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and toxicity of SCH 66336 and gemcitabine in patients with advanced transitional cell carcinoma of the urinary tract.
* Determine the time to progression and objective response rate of this treatment regimen in these patients.
* Assess the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and oral SCH 66336 twice a day (starting on day 2 of the first course, and starting on day 1 of all subsequent courses). Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks until disease progression.

PROJECTED ACCRUAL: A total of 7-31 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or unresectable primary transitional cell carcinoma of the urinary tract, including bladder, ureter, and renal pelvis
* At least one measurable lesion

  * 20 mm or greater by conventional techniques OR
  * 10 mm or greater by spiral CT scan
* Must have received one (and only one) prior chemotherapy regimen for advanced or metastatic disease
* No clinical signs of brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase and transaminases no greater than 2.5 times ULN (no greater than 5 times ULN with liver metastases)

Renal:

* Creatinine no greater than 1.7 mg/dL

Cardiovascular:

* Normal cardiac function
* No ischemic heart disease within the past 6 months
* Normal 12 lead ECG

Other:

* No prior gastrectomy or any gastrointestinal disease that may impair absorption of SCH 66336
* No unstable systemic disease
* No active uncontrolled infection
* No psychological, familial, sociological, or geographical condition that would preclude study
* No prior or concurrent other malignancy except cone biopsied carcinoma in situ of the cervix or adequately treated basal or squamous cell skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No prior farnesyl protein transferase inhibitors or gemcitabine

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* At least 2 weeks since prior major surgery

Other:

* No other concurrent anticancer agents
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2000-06; Primary Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald De Wit, MD, PhD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center; Pieter H. M. de Mulder, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen; Godefridus Peters, PhD, Study Chair — Free University Medical Center
Locations (1):
- University Medical Center Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Result] Theodore C, Geoffrois L, Vermorken JB, Caponigro F, Fiedler W, Chollet P, Ravaud A, Peters GJ, de Balincourt C, Lacombe D, Fumoleau P. Multicentre EORTC study 16997: feasibility and phase II trial of farnesyl transferase inhibitor & gemcitabine combination in salvage treatment of advanced urothelial tract cancers. Eur J Cancer. 2005 May;41(8):1150-7. doi: 10.1016/j.ejca.2005.02.015. PMID 15911238